CLINICAL TRIAL: NCT00058552
Title: A Phase II, Open-label, Multicenter Study to Evaluate the Effect of Tumor-based HER2 Activation on the Efficacy of rhuMAb 2C4 (Pertuzumab) in Subjects With Advanced, Refractory or Recurrent Ovarian Cancer
Brief Title: A Study to Evaluate the Effect of HER2 Activation on rhuMAb 2C4 (Pertuzumab) in Subjects With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: TOC2689g; NCT00070408 (obsolete NCT alias)
Record Dates: First submitted 2003-04-08; First posted 2003-04-09 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Ovarian Cancer
Keywords: Advanced, refractory, or recurrent ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pertuzumab

INTERVENTIONS:
Drug: Pertuzumab (rhuMAb 2C4)

SUMMARY:
The purpose of this study is to determine if the study drug pertuzumab is effective in treating patients with advanced ovarian cancer that is refractory to, or has recurred following, prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Willingness to undergo tumor biopsy and disease that is amenable to biopsy (Cohort 1 only)
* Age >=18 years old
* Advanced, histologically documented carcinoma of the ovary
* Measurable disease with at least one lesion that can be accurately measured per RECIST in at least one dimension (longest dimension recorded). Each lesion must be >=20 mm when measured by conventional techniques, including palpation, plain X-ray, CT, and MRI, or >=10 mm when measured by spiral CT.
* Or, clinically or radiologically detectable disease (e.g., ascites, peritoneal deposits, mesenteric thickening or lesions that do not fulfill RECIST for measurable disease). In addition, the subject must have two consecutive pre-treatment CA 125 levels that are both greater than 2× the institutional upper limit of normal (ULN) and >=40 IU/mL, taken at least 1 week and not more than 3 months apart. The second of the two measurements of CA 125 level should not be drawn within 28 days following the screening biopsy. The later value must be within 2 weeks of starting rhuMAb 2C4 treatment.
* One or more prior platinum-based chemotherapeutic regimens for the management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound
* Life expectancy >=12 weeks
* ECOG performance status 0 or 1
* Use of an effective means of contraception (for women of childbearing potential)
* Granulocyte count >=1500/uL, platelet count of >=75,000/uL, and hemoglobin >=9 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors; darbopoeitin [Aranesp] is permitted)
* Serum bilirubin <=1.5× the ULN and alkaline phosphatase, AST, and ALT <=2.5× ULN (ALT, AST, and alkaline phosphatase <=5× ULN for subjects with liver metastases)
* Serum creatinine <=1.5× ULN
* International normalized ratio (INR) <1.5 and activated partial thromboplastin time (aPTT) <1.5 ULN (except for subjects receiving warfarin)

Exclusion Criteria:

* Prior treatment with experimental anti-cancer agents within 4 weeks prior to Day 1 (the day on which the first rhuMAb 2C4 infusion is administered)
* Prior treatment with HER pathway inhibitors (e.g., Herceptin [Trastuzumab], Iressa [gefitinib], Tarceva [erlotinib hydrochloride], C225, CI1033, and TAK165)
* History or clinical evidence of central nervous system or brain metastases
* Ejection fraction, determined by ECHO, <50%
* Uncontrolled hypercalcemia (>11.5 mg/dL)
* Prior exposure to doxorubicin or liposomal doxorubicin >360 mg/m2 , mitoxantrone >120 mg/m2 , or idarubicin >90 mg/m2
* History of other malignancies within 5 years of Day 1 except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, or basal or squamous cell skin cancer
* History of serious systemic disease, including active infection, uncontrolled hypertension (diastolic blood pressure >100 mmHg on two consecutive occasions), unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation, paroxysmal supraventricular tachycardia, or controlled hypertension are eligible)
* Ongoing liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus infection
* Pregnancy or lactation
* Major surgery or significant traumatic injury within 3 weeks prior to Day 1 with the exception of tumor biopsy for the purposes of the study
* Inability to comply with study and follow-up procedures
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Pertuzumab 420 mg: Participants in this group received pertuzumab intravenous (IV) infusion at a loading dose of 840 milligrams (mg) for Cycle 1 (1 Cycle equals to [=] 3 Weeks), followed by 420 mg for Cycles 2 and beyond, up to 1 year (17 cycles) or until disease progression.
- Pertuzumab 1050 mg: Participants in this group received 1050 mg of pertuzumab IV infusion at each cycle (1 Cycle = 3 Weeks) up to 1 year (17 cycles) or until disease progression.
Period: Overall Study
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Started | 65 | 64
Completed | 0 | 2
Not Completed | 65 | 62
Not completed — Died prior to receiving treatment | 4 | 2
Not completed — Disease progression | 52 | 44
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Physician Decision | 2 | 5
Not completed — Clinical disease progression | 0 | 4

BASELINE CHARACTERISTICS:
Population: All the participants who received at least 1 dose of study drug were included in the analysis.
Groups:
- Pertuzumab 420 mg: Participants in this group received pertuzumab IV infusion at a loading dose of 840 mg for Cycle 1 (1 Cycle = 3 Weeks), followed by 420 mg for Cycles 2 and beyond, up to 1 year (17 cycles) or until disease progression.
- Total: Total of all reporting groups
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.9) | 56.5 (11.2) | 57.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 62 | 123
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Response of Complete Response (CR) or Partial Response (PR) Determined by Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 or Cancer Antigen 125 (CA-125) Changes
Description: Response by tumor measurement occurred if there was documented and confirmed CR or PR determined by 2 consecutive investigator assessments that were at least 28 days apart. Response was assessed by either the RECIST v 1.1 or by CA-125 changes, based on measurable or non-measurable disease at baseline. Per RECIST v 1.1 (for measurable disease), CR: disappearance of all target and non-target lesions and normalization of tumor marker level; PR: at least a 30 percent (%) decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Per CA-125 changes (for non-measurable disease), CR: decrease in the CA-125 to within the normal limits and less than (<) 40 international units per milliliter (IU/mL) and no clinical or radiological evidence of disease, PR: a greater than (>) 50 percent (%) decrease in CA-125 values from baseline, and no clinical or radiological evidence of new lesions.
Time Frame: Screening and prior to infusion at Cycles 3, 5, 7, 9, 13, and 17 and at follow-up (30 days after the last dose of pertuzumab)
Population: Efficacy Analysis Population: All participants who received at least 1 dose of study drug and either underwent at least one postbaseline assessment of response or died within 30 days after the last study treatment before any evaluation of response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 55 | 62
percentage of participants | 3.6 [0.7 to 11.8] | 4.8 [1.3 to 12.9]

2. Secondary Outcome: Percentage of Participants With Disease Progression or Death (Progression Free Survival [PFS])
Description: PFS was defined as the time from the first day of study drug treatment to the time of documented disease progression or death, whichever came first. Participants who were lost to follow-up or who had not progressed at the time of study completion or early termination were censored at the date of last tumor assessment. The percentage of participants experiencing disease progression or death was calculated as the number of participants with event divided by the number of participants analyzed, multiplied by 100.
Time Frame: as for outcome 1
Population: Efficacy Analysis Population. Six participants in pertuzumab 420 mg treatment arm and 15 participants in pertuzumab 1050 mg treatment arm were censored for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 55 | 62
percentage of participants | 89.1 | 75.8

3. Secondary Outcome: Median Time of PFS
Description: PFS was defined as the time from the first day of study drug treatment to the time of documented disease progression or death, whichever came first. Participants who were lost to follow-up or who had not progressed at the time of study completion or early termination were censored at the date of last tumor assessment.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 55 | 62
weeks | 7.6 [6.0 to 11.4] | 6.1 [5.9 to 11.4]

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the initial CR or PR to the time of disease progression.
Time Frame: as for outcome 1
Population: Only responders (CR or PR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 2 | 3
weeks | 18.6 [17.9 to 19.4] | 21.1 [13.1 to 29.1]

5. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants experiencing death was calculated as the number of participants with event divided by the number of participants analyzed, multiplied by 100.
Time Frame: Days 1, 8, and 15 of Cycles 1 and 2, Day 1 of Cycles 3-17, follow-up (30 days after the last dose of pertuzumab) and then every 3 months until death or loss to follow-up (up to 5 years)
Population: Efficacy Analysis Population.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 55 | 62
percentage of participants | 69.1 | 46.8

6. Secondary Outcome: Overall Survival
Description: Survival was the interval of time from date of first dose of study medication to date of death at any time. Participants who had not died were censored at the date of last contact when they were known to be alive.
Time Frame: as for outcome 5
Population: Efficacy Analysis Population. Seventeen participants in pertuzumab 420 mg arm and 33 participants in pertuzumab 1050 mg were censored for this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 55 | 62
weeks | 46.7 [30.4 to 66.6] | NA [38.9 to NA] — Data for 33 participants were censored, thus median and confidence interval upper limit were not reached.

7. Secondary Outcome: Kaplan Meier Estimate of Percentage of Participants Who Were Free of Disease Progression at 3, 6, and 12 Months
Description: Per RECIST v 1.1, disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions, and/or unequivocal progression of existing non-target lesions.
Time Frame: 3, 6, and 12 months
Population: Efficacy Analysis Population.
Measure: Number; unit: percentage of participants
Groups:
- Pertuzumab 420 mg: Participants in this group received pertuzumab at a loading dose of 840 mg for Cycle 1, followed by 420 mg for Cycles 2 and beyond, up to 1 year (17 cycles) or until disease progression (1 Cycle = 3 Weeks).
- Pertuzumab 1050 mg: Participants in this group received 1050 mg of pertuzumab at each cycle (1 Cycle = 3 Weeks) up to 1 year (17 cycles) or until disease progression.
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 55 | 62
percentage of participants
  % of participants free from PD at 3 months | 25.5 | 24.2
  % of participants free from PD at 6 months | 7.3 | 6.5
  % of participants free from PD at 12 months | 0.0 | 0.0

ADVERSE EVENTS:
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Serious Adverse Events (participants affected / at risk) | 26/61 | 18/62
Other Adverse Events (participants affected / at risk) | 61/61 | 60/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 420 mg (N=61) | Pertuzumab 1050 mg (N=62)
Small intestinal obstruction (Gastrointestinal disorders) | 8 | 6
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Abdomial pain (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Endocarditis noninfective (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthenia (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Intestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 420 mg (N=61) | Pertuzumab 1050 mg (N=62)
Diarrhoea (Gastrointestinal disorders) | 40 | 45
Abdominal pain (Gastrointestinal disorders) | 25 | 20
Nausea (Gastrointestinal disorders) | 22 | 22
Vomiting (Gastrointestinal disorders) | 22 | 17
Constipation (Gastrointestinal disorders) | 17 | 11
Abdominal distention (Gastrointestinal disorders) | 13 | 8
Dyspepsia (Gastrointestinal disorders) | 6 | 13
Stomatitis (Gastrointestinal disorders) | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 7 | 4
Ascites (Gastrointestinal disorders) | 5 | 3
Abdominal discomfort (Gastrointestinal disorders) | 2 | 5
Haematochezia (Gastrointestinal disorders) | 4 | 2
Fatigue (General disorders) | 21 | 33
Odema peripheral (General disorders) | 13 | 14
Pyrexia (General disorders) | 7 | 4
Asthenia (General disorders) | 8 | 2
Pain (General disorders) | 5 | 3
Chills (General disorders) | 4 | 3
Early satiety (General disorders) | 2 | 4
Oedema (General disorders) | 4 | 1
Mucosal inflammation (General disorders) | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 15 | 12
Dehydration (Metabolism and nutrition disorders) | 12 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 5
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 14 | 16
Pruritis (Skin and subcutaneous tissue disorders) | 8 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 7
Erythema (Skin and subcutaneous tissue disorders) | 4 | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 1
Ejection fraction decreased (Investigations) | 11 | 13
Weight decreased (Investigations) | 10 | 9
Haemoglobin decreased (Investigations) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Headache (Nervous system disorders) | 10 | 6
Dizziness (Nervous system disorders) | 7 | 6
Dysgeusia (Nervous system disorders) | 4 | 2
Paraesthesia (Nervous system disorders) | 4 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Urinary tract infection (Infections and infestations) | 6 | 8
Sinusitis (Infections and infestations) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Rhinitis (Infections and infestations) | 5 | 1
Insomnia (Psychiatric disorders) | 10 | 5
Anxiety (Psychiatric disorders) | 6 | 5
Depression (Psychiatric disorders) | 6 | 2
Anaemia (Blood and lymphatic system disorders) | 9 | 10
Dysuria (Renal and urinary disorders) | 7 | 6
Haematuria (Renal and urinary disorders) | 5 | 2
Tachycardia (Cardiac disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.